CLINICAL TRIAL: NCT00589758
Title: Tissue Doppler Assessment of Right Ventricular Performance in Acute Heeart Failure
Acronym: TARVA
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 06-467
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Diseases
Keywords: Right Ventricle; Echocardiogram; Evaluation of Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Decompensated Heart Failure: Admitted to Heart Failure ICU for acute decompensated heart failure. 2D and 3D echocardiography will be obtained at baseline, 24 -48 hours and 1-2 weeks post discharge.
  Blood and urine will be collected for biomarker evaluation at each timepoint
  Interventions: Diagnostic Test: Echocardiography; Other: Biomarker evaluation

INTERVENTIONS:
Diagnostic Test: Echocardiography — 2D and 3D echocardiography
Other: Biomarker evaluation — Blood and urine collected

SUMMARY:
The primary purpose of this study is to learn if taking pictures of your heart using two dimensional and three dimensional echocardiography in the heart failure intensive care unit can be helpful to understanding how the heart is working.

All research subjects will be adults admitted to the heart failure ICU with acute decompensated heart failure and requiring monitoring of their heart function using a catheter that is placed in the pulmonary artery which is a blood vessel. In this situation, use of the pulmonary artery catheter,or PAC, is considered standard clinical care. It is not a research procedure. The PAC would be used even if you were not participating in this research project.

All research subjects will be evaluated at the time they are admitted to the ICU, 24 to 48 hours after admission to the ICU, and 7 days after leaving the ICU. At all three time points, we will be taking pictures of the heart using the two dimensional and three dimensional echocardiogram.

Additionally, at each time-point, we will collect a blood sample of approximately two and a half tablespoons each time, and a urine sample. We will be testing the sample for biomarkers of heart failure which are proteins and enzymes specifically related to heart function. We will not be conducting any genetic research on the sample. Any extra blood from these research tests will not be saved for future research.

We will also be looking at the data that is collected by the pulmonary artery catheter. The catheter has a sensor on it that measures things like blood flow and pressure in the heart.

At the Day 7 post discharge visit there will be a six minute hall walk so that we can access the distance that you can walk. We will access any symptoms that you may experience. A nurse or physician will monitor the six minute hall walk.

The research information that we collect on you will not be placed in your medical record. The data is for research purposes only.

DETAILED DESCRIPTION:
Study Design This is a single-center, prospective cohort study. The project will be carried out at the Main Campus of the Cleveland Clinic Foundation. Comprehensive transthoracic echocardiography will be performed in the Heart Failure Intensive Care Unit at the Cleveland Clinic Foundation. This is an eight bed intensive care unit dedicated to treating patients with acute clinical issues related to heart failure and is staffed by heart failure specialists, medical officers and nurses specializing in heart failure management.

Therapy will be individualized per patient and will be entirely at the discretion of the patients' cardiologist under the standard of care. Nevertheless, the Heart Failure Intensive Care Unit has standard drug protocols for intravenous vasodilators such as nitroglycerin and sodium nitroprusside, as well as inotropic therapy such as dobutamine and or milrinone, and pressors such as norepinephrine and or vasopressin. Based on the hemodynamic assessment using PAC, diuretics and vasodilators will be the first-line agents, followed by inotropic agents. Oral vasodilators will be instituted following a standard protocol. All medications and their doses will be noted at the time of each echocardiographic evaluation.

The schedule will be as follows:

1. The first echo will be performed within 24 hours of PAC insertion. Preferably at the time of or prior to commencing treatment in the Heart Failure Intensive Care unit.
2. The second echo will be performed 24-72 hours after baseline echo in the Heart Failure Intensive Care unit.
3. The third echo will be performed at the time of the scheduled outpatient visit after hospital discharge. The tests will be performed in the General Clinical Research Center which is an outpatient visit located on the fifth floor of the M building or at Cardiology Desk F-17.

Timeline for individual patients:

Data Extraction

Invasive Hemodynamics:

All patients will have a PAC inserted, usually via right jugular venous approach, for a clinical indication prior to recruitment This is required for inclusion into the study. Data collected at baseline and at the time of second echo will include systolic and diastolic blood pressures, heart rate and rhythm, central venous pressure, systolic and mean pulmonary artery pressures, pulmonary capillary wedge pressure, cardiac output and index by Fick equation, calculated cardiac power, systemic and pulmonary vascular resistance, and transpulmonary gradient. Thermodilution derived RV ejection fraction can also be performed. A dedicated hemodynamic database capturing all the above mentioned variables has already been designed and implemented for routine clinical use in the Heart Failure Intensive Care Unit. Since this is an observational study, it can be performed in concurrent with other clinical trials.

Echocardiographic studies:

All echocardiograms will be performed on an ultrasound machine capable of two dimensional echocardiograms with strain imaging using the GE Vivid 7 machine and three dimensional echocardiograms using the GE Vivid 7 machine or Phillips ultrasound machine.

Each patient will undergo echocardiographic assessment with a standard ultrasound machine equipped with a 3.5 MHz transducer and capable of digital image storage. All echocardiograms will be performed on an ultrasound machine at the bedside, capable of two dimensional echocardiography with strain imaging using GE Vivid 7machine, and three dimensional echocardiography using the GE Vivid 7 machine or Phillips ultrasound machine. The reason for the broad range of study periods is to allow flexibility of performing echocardiography to fit into the patients' treatment plan in the Heart Failure Intensive Care Unit. Our experience in conducting this kind of study in the Heart Failure Intensive Care Unit has led us to believe that having a range of times is often helpful. Patients admitted overnight or in the weekends, without compromising the objectives of the study. Since the objective of the study is to determine the role of serial echocardiographic parameters with or without hemodynamic data in predicting the need for more invasive interventions or correlating with treatment responses to infusions, this design is close to "real-world" logistics and will unlikely affect study results.

Patients will be placed in the left lateral decubitus position. When this is not possible such as when a patient is on a ventilator, modified views will be obtained. Standard parasternal long and short axis as well as standard apical four, three and two chamber views will be obtained. Subcostal images will be acquired when possible. The echocardiogram will include assessment of left and right ventricular systolic and diastolic function and valvular function. Assessment of systolic function will include: left ventricular end-systolic and end-diastolic diameters, left ventricular outflow tract diameter, left ventricular volumes, pulsed Doppler of Left ventricular outflow tract. Biplane left ventricular ejection fraction, stroke volume, cardiac output and index will then be calculated. Right-sided measurements will include, right ventricular end diastolic and systolic areas, pulse wave Doppler of the tricuspid valve. Strain will be acquired in all views along with pulse wave tissue Doppler of left and right ventricular annuli.

Cardiac Biomarkers:

A total of 40cc blood sample collection in plasma (20cc) and serum (20cc) will be collected at each echo study, and will be processed and aliquotted within 2 hours at the GCRC core lab. Biomarkers of interest include: (1) plasma B-type natriuretic peptide at every visit, (2) cardiac troponin T at baseline, (3) high-sensitive C-reactive protein (hsCRP) at baseline, will be sent to the clinical laboratory for analysis. Extra blood will be collected at every visit and stored in -80F freezer for other research-based novel biomarkers, all subject to availability of supplementary external research funding.

Six minute hall walk Standard Six minute hall walk will be performed to assess functional capacity only at the GCRC follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* admission to H-22 with Acute Decompensated Heart Failure
* clinical indication for PAC placement

Exclusion Criteria:

* pericardial constriction or tamponage on echo or by other imaging modality
* status post cardiac transplantation
* inability to provide informed consent or unable or unwilling to follow protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to H22 ICU
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Surrogate marker of hemodynamic responses to therapy. | Admission to ICU - 2 weeks post discharge
  Correlation of peak systolic right ventricular strain with PCWP

CONTACTS AND LOCATIONS:
Overall Officials: James Thomas, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No